CLINICAL TRIAL: NCT03335098
Title: A Phase 2 Study to Evaluate the Efficacy of Bortezomib in Patients With De-novo Waldenstrom's Macroglobulinemia and Lymphoplasmacytic Lymphoma
Brief Title: Study of VTD in Waldenstrom's Macroglobulinemia
Acronym: BOMB-THROW
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Youngil Koh, Assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1605-137-765
Record Dates: First submitted 2017-11-04; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma
Keywords: Waldenstrom's macroglobulinemia; Lymphoplasmacytic lymphoma; Bortezomib; Thalidomide
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone | interventions — Bortezomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Subcutaneous bortezomib 1.3mg/m2 on days 1, 4, 8, and 11 (every 4 weeks, up to 6 cycles) Oral thalidomide 50mg daily on days 1-28 (every 4 weeks, up to 6 cycles) Intravenous or oral dexamethasone 40mg on days 1-4 (every 4 weeks, up to 6 cycles)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Six 4-week cycles
  Other Names: Thalidomide; Dexamethasone

SUMMARY:
This study is a phase 2, single-arm, open-label, multi-institutional trial to evaluate the efficacy of combination therapy of bortezomib, thalidomide, and dexamethasone in patients with newly diagnosed Waldenstrom's macroglobulinemia and lymphoplasmacytic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 or older
* Newly diagnosed Waldenstrom's macroglobulinemia or lymphoplasmacytic lymphoma
* Previously untreated with chemotherapy
* ECOG performance status of 2 or lesser
* Peripheral blood white blood cell count ≥ 3,500/uL
* Peripheral blood neutrophil count ≥ 1,000/uL
* Peripheral blood platelet count ≥ 20,000/uL
* Peripheral blood hemoglobin ≥ 6.0g/dL
* Serum total bilirubin ≤ 2.0 mg/dL
* Serum aspartate aminotransferase ≤ 2.5 x (upper normal limit)
* Serum alanine aminotransferase ≤ 2.5 x (upper normal limit)

Exclusion Criteria:

* Diagnosed with other malignancy within 5 years before enrollment
* Prior hematopoietic stem cell transplantation
* Prior organ transplantation
* Uncontrolled central nervous system involvement
* Congenital immunodeficiency
* Acquired immune deficiency syndrome (AIDS)
* Pregnancy
* Uncontrolled epilepsy
* Uncontrolled psychological disease
* Peripheral neuropathy of grade 3 or higher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | at 3 years
  Overall response rate as per Lugano criteria

SECONDARY OUTCOMES:
Progression-free survival | at 3 years
  Time from enrollment to disease progression or death from any cause
Overall survival | at 3 years
  Time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
IPD regarding participant demographics, study treatment, response, survival, and adverse events will be shared after publishment of the study results.
Time Frame: IPD will be shared after the publication of the study results without time limit.
Access Criteria: IPD will be shared only for the research purpose.